CLINICAL TRIAL: NCT07297550
Title: Phase Ib/II Study to Evaluate Safety and Preliminary Efficacy of the JAK1 Inhibitor Combined With Intensive Immunosuppressive Therapy in Severe Aplastic Anemia
Brief Title: Safety and Efficacy of the JAK1 Inhibitor Combined With Intensive Immunosuppressive Therapy in Severe Aplastic Anemia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Jun Shi, Director of the Red Blood Cell Diseases Center & Director of the Regenerative Medicine Clinic, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025131
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Severe Aplastic Anemia; Refractory Aplastic Anemia; Newly Diagnosed Aplastic Anemia
Keywords: JAK1 inhibitor; Intensive immunosuppressive therapy
MeSH Terms: conditions — Anemia, Aplastic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JAK1 inhibitor (Experimental): Phase Ib:
  Dose escalation follows the "3+3" principle. Participants will receive golidocitinib 150 mg every other day (qod) or 150 mg once daily (qd) for 12 consecutive weeks. Based on the clinical trial data obtained (e.g., safety, maximum tolerated dose), the recommended Phase II dose (RP2D) will be determined following discussion by the SRC.
  Phase II:
  Participants will receive golidocitinib at the RP2D in combination with intensive immunosuppressive therapy for 12 consecutive weeks.
  intensive immunosuppressive therapy regimen:
  * Porcine anti-lymphocyte globulin (pALG): 25 mg/kg/day or Rabbit anti-thymocyte globulin (rATG): 3.0 mg/kg/day × 5 days,
  * Cyclosporine: 3-5 mg/kg/day,
  * Eltrombopag: 15 mg/day.
  Interventions: Drug: Golidocitinib Capsules

INTERVENTIONS:
Drug: Golidocitinib Capsules — In phase Ib, the low-dose cohort will receive golidocitinib 150 mg orally every other day (qod), and the high-dose cohort will receive golidocitinib 150 mg orally once daily (qd).

SUMMARY:
This study is designed as a Phase Ib/II trial. The phase Ib cohort will enroll patients with severe aplastic anemia (SAA) who have failed to respond to intensified immunosuppressive therapy. In contrast, the phase II cohort will include newly diagnosed and treatment-naïve patients with SAA. A Safety Review Committee (SRC), chaired by the principal investigators, will be established to oversee patient safety throughout the study. Suppose the Phase Ib results demonstrate acceptable safety and tolerability. In that case, the data will be submitted to the Ethics Committee for review, and, upon approval, the study will advance to Phase II.

Phase Ib uses a 3+3 dose-escalation design with two cohorts: 150 mg golidocitinib orally every other day (low dose) or once daily (high dose). Phase II is a single-arm trial with Simon's two-stage optimal design.

ELIGIBILITY:
Phase Ib:

Inclusion Criteria:

* According to the Chinese Guidelines for the Diagnosis and Treatment of Aplastic Anemia (2022 Edition) and the Guidelines for the diagnosis and management of adult aplastic anaemia: A British Society for Haematology Guideline (Br J Haematol. 2024; 204: 784-804), the patient is diagnosed with primary acquired AA and meets the diagnostic criteria for SAA.
* Subjects received intensive immunosuppressive therapy combined with a standard-dose TPO receptor agonist for at least 4 months but failed to respond or experienced relapse.
* Unsuitable for or unwilling to undergo allogeneic hematopoietic stem cell transplantation and lacking other superior treatment options.
* Age ≥ 18 years
* ECOG performance status ≤2
* Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

* Presence of any other primary or secondary bone marrow failure syndrome, including but not limited to Fanconi anemia, myelodysplastic syndrome (MDS), clonal cytopenia of undetermined significance, or large granular lymphocytic leukemia.
* Bone marrow reticulin fibrosis ≥ grade 2
* Subjects with a paroxysmal nocturnal hemoglobinuria (PNH) clone ≥ 50% or with evidence of active hemolysis.
* Presence of clonal cytogenetic abnormalities characteristic of MDS, excluding +8, del(20q), and -Y.
* Active infection within 2 weeks before first dosing of the investigational product, including bacterial, viral, or fungal infections (common cold and onychomycosis excluded). Any anti-infective treatment must be completed at least 2 weeks before dosing. History of HIV infection or HIV antibody positive at screening. Positive treponemal antibody for syphilis at screening. Active pulmonary tuberculosis, defined as evidence of active TB on chest imaging or other relevant assessments within 3 months before first dosing or during screening. Active hepatitis at screening, defined as: HBsAg positivity; or HBcAb positivity with HBV DNA ≥ 30 IU/mL; or HCV antibody positivity with detectable HCV RNA.
* Active bleeding involving the gastrointestinal tract, respiratory tract, central nervous system, or other sites.
* History of clinically significant diseases that, in the investigator's judgment, may pose a risk to the participant's safety if enrolled in the study, or may interfere with the assessment of efficacy or safety during the study, including but not limited to: 1. Cardiovascular diseases: history within the past year of acute myocardial infarction or unstable angina, severe arrhythmias (e.g., frequent multifocal ventricular premature beats, ventricular tachycardia, ventricular fibrillation), congestive heart failure, arterial or venous thrombosis, or New York Heart Association (NYHA) class III-IV heart failure. 2. History of psychiatric disorders or presence of severe cerebrovascular disease or cognitive sequelae.
* Treatment with mycophenolate mofetil, tacrolimus, sirolimus, cyclophosphamide, anti-CD52 monoclonal antibody, or other similar therapies within 4 weeks or 5 half-lives of the first dose of the investigational product, whichever is shorter.
* Planned participation in another clinical trial, or prior exposure to investigational products in another clinical trial within 4 weeks or within 5 half-lives of the first dose of the investigational product, whichever is shorter.
* Received a live attenuated vaccine within 4 weeks before the first dose of the investigational product, planned administration of a live attenuated vaccine during the study, or received a COVID-19 vaccine within 7 days before dosing.
* Prior treatment with a JAK inhibitor.
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study; female participants of childbearing potential and male participants whose partners are of childbearing potential who do not agree to use highly effective contraception throughout the study period (from signing the ICF until 6 months after the last dose of the investigational product), or those planning to donate oocytes or sperm during the study.
* Subjects that the investigator believes have other reasons that make them unsuitable for inclusion in this study.

Phase II:

Inclusion Criteria:

* According to the Chinese Guidelines for the Diagnosis and Treatment of Aplastic Anemia (2022 Edition) and the Guidelines for the diagnosis and management of adult aplastic anaemia: A British Society for Haematology Guideline (Br J Haematol. 2024; 204: 784-804), the patient is diagnosed with primary acquired AA and meets the diagnostic criteria for SAA.
* Meets the diagnostic criteria for severe aplastic anemia (Br J Haematol. 2024; 204: 784-804), which require: 1. Bone marrow cellularity less than 25% of normal; if ≥ 25% but < 50%, residual hematopoietic cells must be < 30%. 2. Peripheral blood counts must meet at least two of the following three criteria: Absolute neutrophil count (ANC) < 0.5 × 10^9/L, Absolute reticulocyte count < 60 × 10^9/L, Platelet count (PLT) < 20 × 10^9/L
* Unsuitable for or unwilling to undergo allogeneic hematopoietic stem cell transplantation.
* Age ≥ 18 years
* ECOG performance status ≤2
* Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

* Presence of any other primary or secondary bone marrow failure syndrome, including but not limited to Fanconi anemia, myelodysplastic syndrome (MDS), clonal cytopenia of undetermined significance, or large granular lymphocytic leukemia.
* Bone marrow reticulin fibrosis ≥ grade 2
* Subjects with a paroxysmal nocturnal hemoglobinuria (PNH) clone ≥ 50% or with evidence of active hemolysis.
* Presence of clonal cytogenetic abnormalities characteristic of MDS, excluding +8, del(20q), and -Y.
* Participation in another clinical trial and use of investigational products or medical devices within 30 days prior to the first dose of the investigational product or within 5 half-lives of the investigational product, whichever is longer.
* Prior use of any of the following before the first dose of the investigational product: rabbit anti-thymocyte globulin (rATG) or porcine anti-lymphocyte globulin (pALG); alemtuzumab; or medium- to high-dose cyclophosphamide (≥30-45 mg/kg/day).
* Prior use of standard-dose cyclosporine or standard-dose TPO-RA for more than 1 month before the first dose of the investigational product.
* Bleeding and/or infection that remain uncontrolled despite receiving standard therapy prior to the first dose of the investigational product.
* Active CMV or EBV infection.
* History of, or concurrent presence of: Positive human immunodeficiency virus (HIV) antibody test; Positive hepatitis B surface antigen (HBsAg), or positive hepatitis B core antibody (HBcAb) with HBV DNA above the assay upper limit of quantification.
* Uncontrolled conditions prior to the first dose of the investigational product, including: 1. Hypertension: blood pressure remains uncontrolled despite lifestyle modification and treatment with two or more appropriately dosed, tolerable antihypertensive drugs (including diuretics) for more than 1 month, or requiring four or more antihypertensive drugs for effective control. 2. Severe arrhythmias, such as complete left bundle branch block, atrial fibrillation, or torsades de pointes. 3. Unstable angina. 4. Pulmonary hypertension, defined as estimated pulmonary artery systolic pressure (PASP) ≥ 60 mmHg by echocardiography. 5. Active bleeding involving the gastrointestinal tract, respiratory tract, central nervous system, or other sites.
* Any arterial or venous thrombosis within 1 year prior to the first dose (excluding fully resolved deep or superficial venous thromboembolism), such as myocardial infarction or pulmonary embolism.
* History of other malignancies within 5 years prior to the first dose (excluding cured early-stage tumors such as basal cell or squamous cell skin cancer, early-stage papillary thyroid cancer, superficial bladder cancer, cervical or breast carcinoma in situ, or localized prostate cancer with Gleason score <6).
* Pregnant or breastfeeding.
* Presence of contraindications to rATG, pALG, or cyclosporine.
* Prior treatment with a JAK inhibitor.
* Subjects that the investigator believes have other reasons that make them unsuitable for inclusion in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Within 12 weeks
  This primary outcome measure applies to Phase Ib, and adverse events will be assessed using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Percentage of patients with complete hematological response | Within 3 months post treatment
  This primary outcome measure applies to Phase II, and a complete hematological response (CR) is defined as meeting all of the following criteria: 1) HGB ≥ 100 g/L; 2) PLT ≥ 100 × 10^9/L; 3) ANC ≥ 1.0 × 10^9/L.

IPD SHARING:
Plan to Share IPD: No